CLINICAL TRIAL: NCT04004429
Title: A Double-blind, Multicenter, Two-part, Randomized, Placebo-controlled Study of the Safety, Tolerability, and Efficacy of 4 Weeks Treatment With AP1189 in Early Rheumatoid Arthritis (RA) Patients With Active Joint Disease
Brief Title: A Study of the Safety, Tolerability and Efficacy of Treatment With AP1189 in Early RA Patients With Active Joint Disease
Acronym: BEGIN
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SynAct Pharma Aps (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SynAct-CS002
Record Dates: First submitted 2019-06-26; First posted 2019-07-02 (Actual); Results first posted 2024-07-10 (Actual); Last update posted 2024-07-10 (Actual); Status verified 2024-07

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — N-(3-(1-(2-nitrophenyl)-1H-pyrrol-2-yl)allylidenamino)guanidine

STUDY DESIGN:
Intervention Model Description: Multicenter, two-part, randomized, double-blind, placebo-controlled 4-week study with repeated doses of AP1189
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 50 mg AP1189 (Experimental): 50 mg AP1189. The treatment is a 4 week treatment. Each daily dose will be administered as a suspension, i e. the powder will be added 50 ml water.
  Interventions: Drug: 50 mg AP1189
- 100 mg AP1189 (Experimental): 100 mg AP1189. The treatment is a 4 week treatment. Each daily dose will be administered as a suspension, i e. the powder will be added 50 ml water.
  Interventions: Drug: AP1189
- Placebo (Placebo Comparator): Placebo. The treatment is a 4 week treatment. Each daily dose will be administered as a suspension i e. the powder will be added 50 ml water.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: 50 mg AP1189 — 50 mg AP1189 powder in bottle
  Other Names: AP1189
  Arms: 50 mg AP1189
Drug: AP1189 — 100 mg AP1189 powder in bottle
  Arms: 100 mg AP1189
Drug: Placebo — Placebo powder in bottle
  Arms: Placebo

SUMMARY:
This is a multicenter, two-part, randomized, double-blind, placebo-kontrolled, 4-week study with repeated doses of AP1189. The study population will consist of newly diagnosed subjects with severe active Rheumatoid Arthritis, defined with a Clinical Disease Activity score (CDAI) > 22, who are to start up-titration with methotrexate.

DETAILED DESCRIPTION:
A multicenter, two-part, randomized, double-blind, placebo-kontrolled, 4-week study with repeated doses of AP1189. The study population will consist of newly diagnosed subjects with severe active Rheumatoid Arthritis, defined with a Clinical Disease Activity score (CDAI) > 22, who are to start up-titration with methotrexate.

The study will be conducted in two parts separated by an interim analysis.

Part 1: The subjects will be randomized in a 1:1:1 ratio into: .

* AP1189 dose 50 mg
* AP1189 dose 100 mg
* placebo

INTERIM ANALYSIS

Part 2: All subjects will be randomized into either design 1, 2 or 3 based on data from the interim analysis.

* Design 1: AP1189 dose 50 mg or placebo in a 2:1 ratio
* Design 2: AP1189 dose 100 mg or placebo in a 2:1 ratio
* Design 3: Continue with the same doses as in Part 1

The purpose of this study is to determine the safety and efficacy of 2 doses of AP1189 compared with placebo after 4 weeks of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent has been obtained prior to initiating any study specific procedures
* Male and female subjects, 18 to 85 years of age
* Confirmed diagnosis of RA (Rheumatoid Arthritis) according to the 2010 American College of Rheumatology (ACR)/EULAR RA classification criteria
* Polyarthritis with joint swelling and tenderness of a minimum of three joints out of 68 joints tested
* Candidate for Methotrexate treatment
* Is about to begin treatment with MTX (Methotrexate)
* Tested positive for anti-CCP (Anti-cyclic citrullinated peptide) or RF (Rheumatoid Factor)
* Severe active RA (Clinical Disease Activity Index (CDAI)) > 22) at screening and baseline
* Negative QFG-IT (QuantiFERON-in-Tube test)
* Subjects should be able to complete the PRO (Patient Reported Outcome) questionnaires
* Females of child-bearing potential may only participate if using reliable means of contraception or are post-menopausal. Surgically sterilized women at least 6 months prior to screening
* Females of childbearing potential must have a negative pregnancy test at screening and baseline

Exclusion Criteria:

* Participation in any other study involving investigational drug(s) within 4 weeks prior to study entry
* Major surgery within 8 weeks prior to screening or planned surgery within 1 month following randomization
* Rheumatic autoimmune disease other than RA, including SLE (systemic Lupus Erythematosus), MCTD (Mixed Connective Tissue Disease), scleroderma, polymyositis, or significant systemic involvement secondary to RA. Sjögren syndrome with RA is allowable
* Functional class IV as defined by the ACR Criteria for Classification of Functional Status in RA or wheelchair/bedbound
* Prior history of or current inflammatory joint disease other than RA
* Subjects with fibromyalgia
* Initiation or change in dose for NSAIDs within 2 weeks prior to dosing with the IMP (Investigational Medicinal Product)
* Corticosteroids are prohibited within 2 weeks prior to screening (and during the entire treatment period and until the final visit
* Evidence of serious uncontrolled concomitant cardiovascular, nervous system, pulmonary, renal, hepatic, endocrine, or gastrointestinal disease
* Have prior renal transplant, current renal dialysis or severe renal insufficiency (determined by a derived glomerular filtration rate (GFR) using Cockcroft Gault Formula of ≤30 mL/min/1,73 m2 calculated by the local lab)
* Uncontrolled disease states, such as asthma, psoriasis, or inflammatory bowel disease where flares are commonly treated with oral or parenteral corticosteroids
* Evidence of active malignant disease
* Pregnant women or nursing mothers
* History of alcohol, drug, or chemical abuse within the 6 months prior to screening
* Neuropathies or other painful conditions that might interfere with pain evaluation
* Body weight of >150 kg

Exclusion criteria that only applies for Norway

* Evidence of moderate and/or severe organ dysfunction
* Abnormal chest x-ray (as per the discretion of the investigator
* Evidence of positive hepatitis serology
* Evidence of peptic ulcer disease

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2019-08-26 (Actual); Primary Completion 2021-11-16 (Actual); Study Completion 2021-11-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ellen-Margrethe Hauge, Professor, Principal Investigator — Aarhus University Hospital; Espen A Haavardsholm, Concultant, PhD, Principal Investigator — Diakonhjemmet Hospital
Locations (2):
- Aarhus Universitetshospital, Aarhus, Denmark
- Diakonhjemmet Sykehus, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 50 mg AP1189 | 100 mg AP1189 | Placebo
Started (The number of participants started reflects the total number in the study, i.e. both patients from part 1 and part 2. Data from the individual parts have not been analyzed separately.) | 35 | 36 | 34
Completed | 33 | 34 | 32
Not Completed | 2 | 2 | 2
Not completed — Protocol Violation | 1 | 0 | 0
Not completed — Physician Decision | 0 | 1 | 1
Not completed — Withdrawal by Subject | 1 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 50 mg AP1189 | 100 mg AP1189 | Placebo | Total
Number analyzed (Participants) | 35 | 36 | 34 | 105
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 25 | 26 | 25 | 76
  >=65 years | 10 | 10 | 9 | 29
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 28 | 27 | 82
  Male | 8 | 8 | 7 | 23
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 2 | 2
  Not Hispanic or Latino | 35 | 36 | 32 | 103
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Norway | 2 | 0 | 1 | 3
  Denmark | 13 | 15 | 15 | 43
  Sweden | 3 | 3 | 1 | 7
  Moldova | 8 | 6 | 7 | 21
  Bulgaria | 9 | 12 | 10 | 31

OUTCOME MEASURES:

1. Primary Outcome: Change in Clinical Disease Activity Index (CDAI)
Description: The change in CDAI from severe (CDAI > 22) to moderate (CDAI <= 22) after 4 weeks treatment compared to baseline.
  CDAI is calculated as a sum of:
  * SJC (28): Number of Swollen 28-Joint Count (shoulders, elbows, wrists, MCPs, PIPs including thumb IP, knees);
  * TJC (28): Number of Tender 28-Joint Count (shoulders, elbows, wrists, MCPs, PIPs including thumb IP, knees)
  * PGA: Patient Global Disease Activity (patient's self-assessment of overall RA disease activity on a scale 0-100, where 100 is maximal activity)
  * IGA: Physician's Global Disease Activity (evaluator's assessment of the subject's overall RA disease activity on a scale 0-100, where 100 is maximal activity)
Time Frame: 4 weeks
Population: The number of participants analyzed differs from the overall number of participants. Participants that received rescue medication during the treatment period was excluded from the analyses.
Measure: Count of Participants; unit: Participants
Arm/Group | 50 mg AP1189 | 100 mg AP1189 | Placebo
Number analyzed (Participants) | 29 | 33 | 30
Participants | 18 | 17 | 12

2. Primary Outcome: Change in Clinical Disease Activity Index (CDAI)
Description: The change in CDAI after 4 weeks treatment compared to baseline.
  CDAI is calculated as a sum of:
  * SJC (28): Number of Swollen 28-Joint Count (shoulders, elbows, wrists, MCPs, PIPs including thumb IP, knees);
  * TJC (28): Number of Tender 28-Joint Count (shoulders, elbows, wrists, MCPs, PIPs including thumb IP, knees)
  * PGA: Patient Global Disease Activity (patient's self-assessment of overall RA disease activity on a scale 0-100, where 100 is maximal activity)
  * IGA: Physician's Global Disease Activity (evaluator's assessment of the subject's overall RA disease activity on a scale 0-100, where 100 is maximal activity).
  The CDAI score range is from 0 - 76, whereas a score of:
  ≤2.8 means Remission >2.8 and ≤10 means Low Disease Activity >10 and ≤22 means Moderate Disease Activity >22 means High Disease Activity
  For the purpose of this study, a decrease in CDAI (improvement) is reported as - xx.xx).
Time Frame: 4 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Calculated score
Arm/Group | 50 mg AP1189 | 100 mg AP1189 | Placebo
Number analyzed (Participants) | 29 | 33 | 30
Calculated score | -11.97 (8.74) | -15.52 (12.70) | -9.33 (10.58)

3. Secondary Outcome: ACR (American College of Rheumatology) Response
Description: Proportion of subjects achieving a response assessed by ACR20.
  The ACR response rate ACR20 is defined as ≥20% improvement in swollen and tender joint counts (SJC/TJC) and 3 of the following 5 assessments: Patient's Global Assessment of Disease Activity, Physician's Global Assessment of Disease Activity, Patient's Assessment of Pain, Health Assessment Questionnaire - Disability Index or C-Reactive Protein.
  Proportion in the context of this protocol refers to number of participants.
Time Frame: 4 weeks
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | 50 mg AP1189 | 100 mg AP1189 | Placebo
Number analyzed (Participants) | 29 | 33 | 30
Participants | 11 | 20 | 10

4. Secondary Outcome: ACR (American College of Rheumatology) Response
Description: Proportion of subjects achieving a response assessed by ACR50.
  The ACR response rate ACR50 is defined as ≥50% improvement in swollen and tender joint counts (SJC/TJC) and 3 of the following 5 assessments: Patient's Global Assessment of Disease Activity, Physician's Global Assessment of Disease Activity, Patient's Assessment of Pain, Health Assessment Questionnaire - Disability Index or C-Reactive Protein.
  Proportion in the context of this protocol refers to number of participants.
Time Frame: 4 weeks
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | 50 mg AP1189 | 100 mg AP1189 | Placebo
Number analyzed (Participants) | 29 | 33 | 30
Participants | 2 | 8 | 4

5. Secondary Outcome: ACR (American College of Rheumatology) Response
Description: Proportion of subjects achieving a response assessed by ACR70.
  The ACR response rate ACR70 is defined as ≥70% improvement in swollen and tender joint counts (SJC/TJC) and 3 of the following 5 assessments: Patient's Global Assessment of Disease Activity, Physician's Global Assessment of Disease Activity, Patient's Assessment of Pain, Health Assessment Questionnaire - Disability Index or C-Reactive Protein.
  Proportion in the context of this protocol refers to number of participants.
Time Frame: 4 weeks
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | 50 mg AP1189 | 100 mg AP1189 | Placebo
Number analyzed (Participants) | 29 | 33 | 30
Participants | 0 | 4 | 1

ADVERSE EVENTS:
Time Frame: All Adverse Event (AE)s were collected starting from the time of signed informed consent and until the final visit (End of Study/Early Termination visit) had occurred. Any AE that was ongoing at the final visit was followed until resolution or until four weeks after the study drug administration, whichever came first.
Arm/Group | 50 mg AP1189 | 100 mg AP1189 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/35 | 0/36 | 0/34
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/36 | 0/34
Other Adverse Events (participants affected / at risk) | 14/35 | 16/36 | 12/34
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 50 mg AP1189 (N=35) | 100 mg AP1189 (N=36) | Placebo (N=34)
Alanine aminotransferase increased (Investigations) | 6 (6) | 0 (0) | 3 (3)
Anemia (Blood and lymphatic system disorders) | 2 (2) | 1 (1) | 1 (1)
Arthritis rheumatoid aggravated (Musculoskeletal and connective tissue disorders) | 3 (4) | 2 (4) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 2 (2) | 0 (0) | 2 (2)
Constipation (Gastrointestinal disorders) | 2 (2) | 3 (3) | 0 (0)
Diarrhea (Investigations) | 1 (1) | 2 (2) | 0 (0)
GGT increased (Investigations) | 3 (3) | 0 (0) | 3 (3)
Headache (Nervous system disorders) | 2 (2) | 5 (5) | 0 (0)
Nausea (Gastrointestinal disorders) | 5 (5) | 7 (8) | 7 (7)
Obstipation (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0)
Sore Throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2021-01-14): https://cdn.clinicaltrials.gov/large-docs/29/NCT04004429/Prot_000.pdf
  • Statistical Analysis Plan (2021-11-22): https://cdn.clinicaltrials.gov/large-docs/29/NCT04004429/SAP_001.pdf